CLINICAL TRIAL: NCT00372047
Title: Evaluation of Excessive UV Irradiation on Skin Aging by Multiphoton Laser Imaging and Biophysical Methods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Jena (Other)
Other Study IDs: 1845-08/06
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Skin Aging

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Device: multiphoton laser imaging

SUMMARY:
In this study, test persons with chronic excessive UV radiation and a control group are examined by multiphoton laser imaging and biophysical methods in order to evaluate the dermal fiber network. We expect to observe signs of advanced skin aging in the test group.

ELIGIBILITY:
Inclusion Criteria:

* non smokers
* contraception
* 12 subjects with chronic excessive UV irradiation
* 12 normal subjects

Exclusion Criteria:

* dermatological and other severe disorders
* pregnancy and lactation
* dermatological topical therapy
* internal medication
* cosmetical intervention at test area

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaatz, Dr., Principal Investigator — Dept. of Dermatology, FSU Jena
Locations (1):
- Department of Dermatology, FSU Jena, Jena, Thuringia, Germany